CLINICAL TRIAL: NCT06811714
Title: Comparison of Total Oxidant and Total Antioxidant Status in Breast Milk After Caesarean Section Under General and Regional Anesthesia
Brief Title: Comparison of Oxidants and Antioxidants in Breastmilk Under Different Anesthesia Protocols
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Özlem Ersoy Karka, Assistant Professor, Duzce University
Other Study IDs: drozlemersoy6
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-06

CONDITIONS: Oxidative Stress
Keywords: oxidative stress; cesarean section; anesthesia, general; anesthesia, regional; breastmilk

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Anesthesia: 64 Patients undergoing cesarean section under general anesthesia
- Regional Anesthesia: 64 Patients undergoing cesarean section under regional anesthesia

SUMMARY:
The goal of this observational study is to determine in women undergoing cesarean section if total oxidant status and total antioxidant status in breastmilk taken at the 6th hour postoperatively changes between general and regional anesthetic protocols.

Researchers will compare general anesthesia and regional anesthesia groups to see if total oxidant status and total antioxidant status in breastmilk taken at the 6th hour postoperatively changes.

Participants will provide 2 ml of breastmilk at the 6th postoperative hour.

DETAILED DESCRIPTION:
In recent years, the rate of cesarean delivery in our country has ranged between 46% and 54%. Anesthesiologists only have safety concerns for the patient during routine surgery. In cesarean section operations, all the changes that occur in the mother can affect the fetus. This makes cesarean section operations more special than other surgeries. Cesarean section operations can be performed under general anesthesia and regional anesthesia methods. In recent years, regional anesthesia has been preferred because of its advantages, such as patient's request, consciousness, no need for intubation, no risk of aspiration, no respiratory depression in the newborn, and no uterine atony. However, general anesthesia is also frequently used in emergencies, patient requests, and contraindications to regional anesthesia.

Breast milk is the most appropriate nutritional product for newborns. Only breast milk is recommended for newborns for the first 4-6 months. During the period when infants are breastfed, some drugs used by the mother may pass into breast milk and cause adverse effects in infants. Most of the cases of adverse effects due to drugs passing into breast milk occur in newborns younger than two months, especially in the first month of life. In line with this information, it is known that anesthetic drugs also pass into breast milk. Whether it is general anesthesia or regional anesthesia, anesthetic drugs are excreted into breast milk in minimal doses. However, studies show that the anesthetic drugs that pass into breast milk are at levels that do not cause serious side effects in the baby.

Many risk factors can cause oxidative stress, including alcohol, drugs, environmental pollutants, intense exercise, inflammation, and sepsis. Biological targets most exposed to oxidative damage include enzymes, cell membranes, and DNA. Oxygen radicals have been implicated as an essential cause of mechanisms that can lead to the rapid degradation of proteins. Free radical-induced changes in proteins increase the degradation of enzymes. Oxidative damage to protein products can affect the activity of enzymes, receptors, and transporter proteins. Oxidatively damaged protein products may contain reactive groups that can damage the cell membrane and many cellular functions. Peroxidation of lipids occurs when biological membranes react with unsaturated fatty acids and proceed by radical chain reaction. Oxidative events cause changes in the physical-chemical properties of membranes and thus alter fluidity and permeability, with membranes disintegrating with swelling of intracellular organelles. DNA and RNA are sensitive to oxidative damage. DNA is thought to be the main target, especially in aging and cancer. Oxidative nucleotides such as glycol, thymidine glycol, and 8-hydroxy-2- deoxyguanosine have increased during oxidative damage to DNA by UV radiation or free radical damage. Mitochondrial DNA has been reported to be more susceptible to oxidative damage in many diseases, including cancer.

In the literature review in which we investigated the effects of anesthesia on breast milk, the amount of drugs such as anesthetic agents, narcotic agents, and muscle relaxants in breast milk in the postoperative period was investigated. However, no study has been found to show how oxidative stress parameters change in breast milk due to both the anesthetic technique used and secondary causes (stress, tissue damage, etc.) caused by the operation in a newly operated mother. Our study aimed to compare oxidative stress parameters in breast milk after cesarean section under general anesthesia and regional anesthesia. A comprehensive research evaluating total oxidant/antioxidant systems was not found in our literature review. Therefore, our study will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cesarean section under general or regional anesthesia
* Patients in the I and II risk groups, according to the American Society of Anesthesiologists (ASA) classification

Exclusion Criteria:

* Pregnant women with ASA III and above,
* Pregnant women with gestational DM or hypertension,
* Pregnant women with an indication for Intensive Care Unit (ICU),
* Pregnant women with chronic obstructive pulmonary disease,
* Pregnant women with morbid obesity,
* Pregnant women with a history of liver or kidney disease,
* Pregnant women with coronary artery disease or heart failure,
* Pregnant women with significant anemia (Hg<7).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women undergoing elective cesarean section under general or regional anesthesia in operating rooms of Duzce University Health Research Center
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2025-02-06 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Total oxidant status | Postoperative 24 hours
  Total oxidant status in breastmilk taken at 6th postoperative hour will be measured.
Total antioxidant status | Postoperative 24 hours
  Total antioxidant status in breastmilk taken at the 6th postoperative hour will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Ersoy Karka, Ass. Prof., Principal Investigator — Düzce University Faculty of Medicine
Locations (1):
- Duzce University, Düzce, Düzce, Turkey (Türkiye)